CLINICAL TRIAL: NCT03047421
Title: Influence of Different Methods of Measurement in the Accuracy of DES-OSA and P-SAP Scores
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, Principal Investigator, Astes
Other Study IDs: NC-DTC
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients included: For all patients scheduled for an anesthetic preoperative consultation, a comparison of accuracy of DES-OSA and P-SAP scores with PSG (polysomnography) will be performed.
  Interventions: Diagnostic Test: Comparison of accuracy of DES-OSA and P-SAP scores

INTERVENTIONS:
Diagnostic Test: Comparison of accuracy of DES-OSA and P-SAP scores — Comparison of accuracy of DES-OSA and P-SAP scores with the result of the PSG (polysomnography)

SUMMARY:
DES-OSA and P-SAP scores have been validated to detect OSA (Obstructive Sleep Apnea).

One item of P-SAP and DES-OSA is the measurement of neck circumference. The aim of this study is to compare the influence of different methods of neck circumference measurement in the accuracy of DES-OSA and P-SAP scores to detect OSA.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for an anesthetic preoperative consultation

Exclusion Criteria:

* < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for an anesthetic preoperative consultation
Sampling Method: Non-Probability Sample
Enrollment: 1682 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of DES-OSA | one month
  Accuracy of different values of DES-OSA (due to different measurement of neck circumference) with the result of PSG.
Accuracy of P-SAP | one month
  Accuracy of different values of P-SAP (due to different measurement of neck circumference) with the result of PSG.

CONTACTS AND LOCATIONS:
Overall Officials: Eric DEFLANDRE, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc of Bouge, Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No